CLINICAL TRIAL: NCT00780364
Title: Sour Taste and Cold Temperature Effects on Pharyngeal Transit Time After Ischemic Stroke:Anatomic and Functional Bases.
Brief Title: Sour Taste and Cold Temperature in Dysphagia
Status: Terminated | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Principal Investigator, Paula Cristina Cola, PhD, UPECLIN HC FM Botucatu Unesp
Other Study IDs: upeclin/HC/FMB-Unesp-18
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2012-06

CONDITIONS: Stroke
Keywords: stroke; sour taste; cold temperature; pharyngeal swallowing
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective is to establish the effect of sour taste and cold temperature on the pharyngeal swallowing transit time after ischemic hemisphere stroke.

DETAILED DESCRIPTION:
Over the past decade there were many studies over normal and pathological swallowing that discuss the influence of taste and temperature. Nevertheless there were many questions on the issue that remains to be solved, including the hemispheric lateralization of lesions dysphagic patients remains also to be fully understood.Swallowing disorder is defined as oropharyngeal dysphagia in presence of alterations in any phase of the complex swallowing dynamics. It could be congenital or acquired, affecting nutritional aspects, hydration, lung function and the individual's social integration [1]. Stroke, has a high incidence among neurological diseases, and cause disturbs on swallowing dynamics presenting signs of dysphagia in at least 50% of cases.A study that analyzed swallowing dynamics by videofluoroscopy in individuals with history of one or more stroke episodes with oropharyngeal dysphagia shows shorter pharyngeal and oropharyngeal transit times with cold stimulus than without them. Other study of heterogeneous neurological diseases such as cerebral palsy, brain trauma, stroke, and Alzheimer's disease, concluded that sour taste improved swallowing, minimizing laryngotracheal penetration and aspiration in individuals with neurological damaged. Chen et al. in an analysis of 42 healthy individuals with several taste bolus found that awareness and arousal could also influence the swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke

Exclusion Criteria:

* instability clinic

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in hospital
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Sour Taste and Cold Temperature in Dysphagia | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Paula C Cola, master, Principal Investigator — São Paulo State University
Locations (1):
- Sao Paulo State University, Botucatu, São Paulo, Brazil